CLINICAL TRIAL: NCT05754307
Title: A "Closed" Surgical Technique for the Treatment of Residual Periodontal Pockets vs Access Flap Utilizing Papilla Preservation Techniques. A Randomized Controlled Trial
Brief Title: A Closed Surgical Technique vs Papilla Preservation Techniques
Acronym: CST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danae A. Apatzidou (Other)
Responsible Party: Sponsor-Investigator, Danae A. Apatzidou, Associate Professor, Aristotle University Of Thessaloniki
Organization: Aristotle University Of Thessaloniki (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AUTh 179/30-11-2022
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Periodontitis
Keywords: interdental periodontal defect; periodontal surgery; papilla preservation; tunnelling technique; closed surgical technique
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Randomised controlled clinical trial having 2 parallel intervention arms for surgical treatment (step 3) of interproximal residual defects (PPD≥6mm and BoP)
Who Masked: Participant, Outcomes Assessor
Masking Description: Treatment is disclosed to the examiner after all data have been collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control surgical technique (Active Comparator): Intrasulcular incisions at the teeth adjacent to the defect, using the simplified papilla preservation technique (SPPT) or modified papilla preservation technique (MPPT). Granulation tissue is excised and debridement via hand and power-driven instruments follows. Flaps are repositioned and papilla are sutured with horizontal internal mattress doubled by a single interrupted interdental suture.
  Interventions: Procedure: Access Flap
- Test surgical technique (Experimental): Strictly intrasulcular incisions are performed at the teeth adjacent to the defect (mid-buccal to mid-lingual) without incising the interdental papilla. Full thickness gingival flaps, at the base of the papilla, which is retained intact, are elevated in a "closed"-tunneling manner, granting access to the interdental osseous defect. Debridement is performed via power-driven tips and mini curettes, without intentional excising the granulation tissue that lines the osseous defect. Flaps are repositioned by gentle pressure and suturing is not required.
  Interventions: Procedure: Closed Surgical Technique

INTERVENTIONS:
Procedure: Access Flap — Intrasulcular incisions at the teeth adjacent to the defect, using the simplified papilla preservation technique (SPPT) or modified papilla preservation technique (MPPT). Granulation tissue is excised and debridement via hand and power-driven instruments follows. Flaps are repositioned and papilla are sutured with horizontal internal mattress doubled by a single interrupted interdental suture.
  Arms: Control surgical technique
Procedure: Closed Surgical Technique — Strictly intrasulcular incisions are performed at the teeth adjacent to the defect (mid-buccal to mid-lingual) without incising the interdental papilla. Full thickness gingival flaps, at the base of the papilla, which is retained intact, are elevated in a "closed"-tunneling manner, granting access to the interdental osseous defect. Debridement is performed via power-driven tips and mini curettes, without intentionally excising the granulation tissue that lines the osseous defect. Flaps are repositioned by gentle pressure and suturing is not required.
  Arms: Test surgical technique

SUMMARY:
A pioneer periodontal surgical approach employing the closed surgical technique (CST) has been designed to gain access to isolated interdental periodontal defects and retain the soft-tissue architecture. This technique is based on a modified tunnelling technique to retract full-thickness gingival flaps from the osseous defect in a closed manner retaining intact the interproximal papilla thus, suturing is not required. A randomised controlled clinical trial will determine the efficacy of the CST versus the access flap employing papilla preservation techniques over a period of 6 months.

DETAILED DESCRIPTION:
This randomised controlled clinical trial will compare the CST over the access flap employing papilla preservation techniques to treat isolated interdental defects in terms of gain in clinical attachment levels, radiographic evidence of bone apposition and local reduction of pro-inflammatory cytokines over a period of 6 months.

1. First visit - initial examination - at least 3 months after initial non-surgical periodontal treatment (Step 1, 2) Update general and dental history Screening of subjects for suitability; Consent form; Randomization of suitable subjects Intra-oral photography Full-mouth charting: Probing pocket depth (PPD), Clinical Attachment Level (CAL), Plaque Index (PI), Bleeding on Probing (BoP), Gingival Recession (Rec) Oral hygiene instructions (soft toothbrush, modified Bass, interdental cleaning) Full mouth supragingival scaling
2. Second visit - Baseline - T0 Collection of Gingival Crevice Fluid (GCF) using sterilized paper strips Radiographic examination of the site (Long-cone paralleling technique using a digital sensor attached to a custom-made silicone bite block for reproducible radiographs) Periodontal site-selected clinical assessment Periodontal surgery (control: access flap with papilla preservation techniques or test: the CST) under local anaesthesia Modification of oral hygiene instructions; post-operative instructions Intra-oral photography
3. Third visit - T1 (2 weeks post-operatively) Suture removal (only in control group) Wound healing visual monitoring by the Early Healing Index (1-5) Oral hygiene instructions Intra-oral photography Questionnaire for subjective feelings and satisfaction
4. Fourth visit - T2 (6 weeks post-operatively) Oral hygiene instructions Intra-oral photography
5. Fifth visit - T3 - Re-evaluation (6 months post-operatively) GCF collection using sterilized paper strips Periodontal full-mouth charting Site-selected periodontal clinical assessment; Probing Pocket depth (PPD), Clinical Attachment Level (CAL), Plaque Index (PI), Bleeding on Probing (BoP), Gingival Recession (Rec Radiographic examination of the site Oral hygiene instructions Intra-oral photography

ELIGIBILITY:
Inclusion Criteria:

* Systematically healthy subjects, not having consumed antibiotics 3 months before surgical periodontal treatment (baseline)
* Smokers <5 cig/day, former smokers or no smokers
* Periodontal patients fulfilling non surgical initial periodontal treatment at least 3 months before surgical periodontal treatment (baseline day) and presenting at least one residual pocket with PPD and CAL ≥6mm and bleeding on probing, located interproximally with intrerdental site ≥2mm.
* Compliant patients presenting high standards of oral hygiene (full mouth Plaque Index <20%) strictly susceptible in Supportive Periodontal Treatment

Exclusion Criteria:

* Untreated active periodontal inflammation
* Poorly controlled systematic diseases
* Disorders compromise wound healing
* Bisphosphonate medications
* Patients under radiotherapy or chemotherapy
* Drug-indused gingival hyperplasia
* Pregnancy or lactation
* Poor compliance during steps 1 and 2 of cause-related periodontal treatment
* Compromised oral hygiene (full mouth Plaque Index >30%), circumferential bone defect or narrow intrerdental site ≤2mm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical Attachment Level | baseline to 6 months
  Determined by a manual periodontal probe(Hu-Friedy XP-23/QW) by a single examiner at the nearest of 1mm
Cementoenamel junction to Bottom of the defect | baseline to 6 months
  Determined on standardised periapical radiographs obtained by the long cone parallel technique

SECONDARY OUTCOMES:
Probing Pocket Depth | baseline to 6 months
  Determined by a manual periodontal probe
Recession | baseline to 6 months
  Determined by a manual periodontal probe
Levels of proinflammatory cytokines | baseline to 6 months
  Determined by ELISA in GCF
Bleeding on Probing | baseline to 6 months
  Determined by a manual periodontal probe
Patient satisfaction and perception | 2 weeks following surery
  Determined on questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Danae Apatzidou, Associate Professor, Study Director — School of dentistry
Locations (1):
- Dental School, Aristotle University, Dept of Preventive Dentistry, Periodontology and Implant Biology, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No
Overall data but not on an individual basis will be disclosed and shared

REFERENCES:
- [Background] Apatzidou DA, Nile C, Bakopoulou A, Konstantinidis A, Lappin DF. Stem cell-like populations and immunoregulatory molecules in periodontal granulation tissue. J Periodontal Res. 2018 Aug;53(4):610-621. doi: 10.1111/jre.12551. Epub 2018 Apr 23. PMID 29687448
- [Background] Apatzidou DA. A pionner surgical technique for isolated periodontal defects by "closed" retraction of the papilla' Front. Dent. Med. (2022) 3:956601. doiQ 10.3389
- [Background] Cortellini P, Prato GP, Tonetti MS. The modified papilla preservation technique. A new surgical approach for interproximal regenerative procedures. J Periodontol. 1995 Apr;66(4):261-6. doi: 10.1902/jop.1995.66.4.261. PMID 7782979
- [Background] Cortellini P, Prato GP, Tonetti MS. The simplified papilla preservation flap. A novel surgical approach for the management of soft tissues in regenerative procedures. Int J Periodontics Restorative Dent. 1999 Dec;19(6):589-99. PMID 10815597
- [Background] Cortellini P, Tonetti MS. A minimally invasive surgical technique with an enamel matrix derivative in the regenerative treatment of intra-bony defects: a novel approach to limit morbidity. J Clin Periodontol. 2007 Jan;34(1):87-93. doi: 10.1111/j.1600-051X.2006.01020.x. PMID 17243998
- [Background] Apatzidou DA, Bakopoulou AA, Kouzi-Koliakou K, Karagiannis V, Konstantinidis A. A tissue-engineered biocomplex for periodontal reconstruction. A proof-of-principle randomized clinical study. J Clin Periodontol. 2021 Aug;48(8):1111-1125. doi: 10.1111/jcpe.13474. Epub 2021 May 14. PMID 33899259